CLINICAL TRIAL: NCT02515552
Title: Web-Based Program for Symptom Management in Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Collinge and Associates, Inc. (Other)
Responsible Party: Principal Investigator, William Collinge, PhD, President, Collinge and Associates, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: FM Wellness Project
Record Dates: First submitted 2015-07-29; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All applicants (Other): Study applicants who consented and completed the application to participate in the Fibromyalgia Wellness Project. From that point forward all subjects used the intervention program to at whatever frequency they chose voluntarily. It was recommended subjects complete a SMARTLog at least three times per week for at least three months.
  Interventions: Behavioral: The Fibromyalgia Wellness Project

INTERVENTIONS:
Behavioral: The Fibromyalgia Wellness Project — Web-based symptom and behavior self-monitoring program with automated feedback derived from the user's personal data. A personal informatics approach is used involving proprietary within-subject statistical analysis procedures to determine user feedback that provides behavioral guidance based on statistically significant change in symptom levels associated with specific user behavior and self-management strategies.

SUMMARY:
Fibromyalgia is a complex chronic illness affecting 6-12 million Americans. Self-management strategies play a key role in reducing symptoms and maintaining functioning. The proposed project offers a web-based self management tool that enables FM sufferers to identify significant linkages between their personal symptom levels and their personal self-management efforts over time in order to plan their own optimal approach to disease management.

DETAILED DESCRIPTION:
This Phase II project will complete development of the SMART (Self-Monitoring and Review Tool) Log program for symptom management and health promotion in FM and evaluate its efficacy in a large web-based trial that will closely emulate its planned application in Phase III. The SMARTLog program is an interactive web-based self-monitoring and feedback intervention that employs proprietary statistical analysis procedures to give the user personally optimized guidance on behavioral, lifestyle and coping strategies that yield effective symptom reduction for that individual. The program incorporates longitudinal collection and analysis of the individual's self-monitoring data followed by delivery of personalized feedback derived from those same personal data. The program helps FM sufferers discover and monitor linkages between specific personal health-related behaviors and management strategies and their symptom levels over time. Feasibility was demonstrated in Phase I by very high retention rates, ratings of satisfaction and perceived relevance, evidence of impact of utilization on improved well-being over the use period, and qualitative data indicating strong interest in continuation with the program.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported presence of fibromyalgia

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 883 (Actual)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change in daily symptom Levels | Baseline to user-defined end date (variable time series design) up to 9 months
  Change in Likert-scaled (0-10) daily symptom severity levels on the SMARTLog tracking instrument. Daily reported levels over multiple days are aggregated to calculate trends over the user-defined reporting period.

SECONDARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire scores | Baseline to user-defined end date (variable time series design) up to 9 months
Change in Self-Efficacy for Chronic Disease Scale scores | Baseline to user-defined end date (variable time series design) up to 9 months
Change in SF12 scores | Baseline to user-defined end date (variable time series design) up to 9 months
Change in Multi-dimensional Health Locus of Control Scale scores | Baseline to user-defined end date (variable time series design) up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: William B Collinge, PhD, MPH, Principal Investigator — Collinge and Associates, Inc.
Locations (1):
- Collinge and Associates, Inc., Eugene, Oregon, United States

REFERENCES:
- [Result] Collinge W, Yarnold P, Soltysik R. Fibromyalgia Symptom Reduction by Online Behavioral Self-monitoring, Longitudinal Single Subject Analysis and Automated Delivery of Individualized Guidance. N Am J Med Sci. 2013 Sep;5(9):546-53. doi: 10.4103/1947-2714.118920. PMID 24251273
- [Derived] Collinge W, Soltysik R, Yarnold P. Fibromyalgia Impact Reduction Using Online Personal Health Informatics: Longitudinal Observational Study. J Med Internet Res. 2020 Apr 7;22(4):e15819. doi: 10.2196/15819. PMID 32131045
- See also: Results article online (open access) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3818828/